CLINICAL TRIAL: NCT02909790
Title: A RandomizEd DoUble Blinded ControllEd Study to Evaluate the Safety and Effectiveness of the CURVE Low Level Laser Therapy (LLLT) for Circumference Reduction of the Waistline.
Brief Title: Study Safety and Effectiveness of CURVE Laser Therapy for Circumference Reduction of the Waistline.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yolo Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCSP-2016- CURVE
Record Dates: First submitted 2016-09-16; First posted 2016-09-21 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Injury to Subcutaneous Tissue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CURVE LLLT treatment (Experimental): Up to 20 subjects are randomly selected to receive Curve Low Level Laser Therapy
  Interventions: Device: Curve Low Level Laser Therapy
- SHAM device treatment (Sham Comparator): Up to 20 subjects assigned to the sham group will be treated with a device that is designed to have the same physical appearance as the treatment group, except that the interlock fuse (grey fuse holder back of device) will be removed prior to treatment. The laser screen will still be active and show to the subject that the treatment time will still be counting down, but will not activate lasers in the treatment paddles
  Interventions: Device: Curve Low Level Laser Therapy

INTERVENTIONS:
Device: Curve Low Level Laser Therapy — Subjects assigned to the treatment group will be treated with 4 multi-paddle low-level diode laser consisting of 8 independent diode laser heads per treatment paddle, each emitting 630-680nm (red) laser light with each diode generating 40mW output ("CURVE" Laser - manufactured by YOLO Medical Inc.).

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of the CURVE Low-Level Laser Therapy for circumference reduction of the waistline.

DETAILED DESCRIPTION:
This study involves research to obtain information on the CURVE. In recent years Low Level Laser therapy devices have grown in popularity due to increased scientific understanding of their mechanism of action, published research, and patients demand for more non-invasive procedures in body contour and fat reduction. LLL are widely used in health clinics, medical spas and in aesthetic medicine in the treatment of cellulite and for inflammatory conditions such as carpal tunnel syndrome. This study will further evaluate the effectiveness of low-level laser treatments without the extraction of adipose tissue using liposuction or in combination with other treatment modalities.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is an adult ≥ 18 years old and <65 years of age
2. Subject has maintained a stable weight for the past 6 months (variation no greater than 10 lbs. from "usual weight").
3. Subject is willing to maintain current diet and exercise regimen for the duration of study.
4. Subject is willing and able to provide written informed consent.
5. Subject is willing to return for all scheduled and required visits.
6. Subject is willing to comply with post-laser treatment cardiovascular exercise.
7. Subject is willing to comply with food and fluid requirements pre-treatment and post-treatment.

Exclusion Criteria:

1. Subject is on an active weight control regimen.
2. Subject has a pacemaker.
3. Subject has a history of epilepsy.
4. Subject has a history of any type of cancer, including skin cancer.
5. Subject had a prior surgical intervention for body sculpting/weight loss such as liposuction, abdominoplasty, gastroplasty, lap band surgery, etc.
6. Subject has a medical, physical, or other contraindications for body sculpting/weight loss.
7. Subject has an active infection, wound or other external trauma to the areas to be treated with the laser.
8. Subject is pregnant, breast feeding, or planning pregnancy prior to study end.
9. Subject is participating in any treatment other than the study procedure (existing or new) to promote body contouring and/or weight loss during the course of study participation.
10. Subject is participating in another research study of a device, medication, biologic, or other agent within 30 days or could, in the opinion of the investigator, affect the results of this study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Reduction of girth measurements for the waistline after successful completion of the three (3) week study procedure. | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Haneef Alibhai, MD, Principal Investigator — UBC Faculty of Medicine

IPD SHARING:
Plan to Share IPD: Undecided